CLINICAL TRIAL: NCT06099314
Title: A Real-world Study of Fruquintinib in the Cross-line Treatment of Refractory mCRC
Brief Title: Fruquintinib in the Cross-line Treatment of Refractory mCRC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Zhenyu Lin, associate chief physician, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Other Study IDs: HMPL-013-C2-CRC05
Record Dates: First submitted 2023-10-17; First posted 2023-10-25 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2023-10

CONDITIONS: Fruquintinib; Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Fruquintinib Rechallenge: 1. third-line treatment with fruquintinib combined with PD-1 inhibitors
  2. fourth-line treatment with fruquintinib combined with TAS-102
  Interventions: Drug: Fruquintinib+PD-1 inhibitors; Drug: Fruquintinib+TAS-102

INTERVENTIONS:
Drug: Fruquintinib+PD-1 inhibitors — Third-line treatment with fruquintinib combined with PD-1 inhibitors. Fruquintinib: 5mg,Oral once daily,2 weeks on/1 week off,Q3W； PD-1 inhibitor：for example, Sintilimab,iv,200mg, Q3W.
Drug: Fruquintinib+TAS-102 — Fourth-line treatment with fruquintinib combined with TAS-102 . Fruquintinib: 3-5mg(Depending on the patient's physical condition), Oral once daily,3 weeks on/1 week off,Q4W； TAS-102:orally, 35mg/m2 twice daily (maximum dose 80mg in a single dose) for days 1-5, repeated every 14 days.

SUMMARY:
This is a real-world study. Patients with metastatic colorectal cancer who have progressed (PD) after third-line treatment with fruquintinib combined with PD-1 inhibitors will receive fruquintinib combined with TAS-102 as fourth-line therapy. The objective of this study was to observe the efficacy and safety of cross-line（from third to fourth line）treatment with fruquinitinib.

DETAILED DESCRIPTION:
This is a real-world study. Patients with metastatic colorectal cancer confirmed by histopathology had previously received 2-line system therapy with fluorouracil, oxaliplatin, irinotecan, anti-VEGF, anti-EGFR (RAS and BRAF wild type) (treatment with anti-VEGF-TKI is not allowed), and had received fruquinitinib combined with PD-1 inhibitors for third-line treatment. After progression (PD) (confirmed by RECIST 1.1 ), fruquinitinib combined with TAS-102 as fourth-line therapy was received. The primary endpoint was observation the overall survival (OS) of fourth-line treatment of mCRC with fruquinitinib and TAS-102. The study objective is to explore the possibility of cross-line rechallenge of fruquinitinib.

ELIGIBILITY:
Inclusion Criteria:

-

To be enrolled in this study, patients must meet all of the following criteria:

1. Age ≥18 years, ≤75 years;
2. No gender limitation;
3. Patients with metastatic colorectal cancer confirmed by histopathology had previously received 2-line system therapy with fluorouracil, oxaliplatin, irinotecan, anti-VEGF, anti-EGFR (RAS and BRAF wild type) (treatment with anti-VEGF-TKI is not allowed), and had received fruquinitinib combined with PD-1 inhibitors for third-line treatment. After progression (PD) (confirmed by RECIST 1.1 ), fruquinitinib combined with TAS-102 as fourth-line therapy was received.
4. Expected survival ≥12 weeks
5. Must have at least one measurable lesion (RECIST1.1).
6. Full organ and bone marrow function.

Exclusion Criteria:

-

Patients will not be admitted to the study if they meet any of the following criteria:

1. Patients with contraindications to study drugs (fruquinitinib, PD-1 inhibitor, TAS-102);
2. allergic to the investigational drug or any of its adjuncts;
3. There are other non-investigational drugs during third-line and fourth-line treatment;
4. Pregnant or lactating female subjects;
5. Patients with a large number of pleural effusion or ascites requiring drainage;
6. Patients considered unsuitable for inclusion in this study by the investigators.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with metastatic colorectal cancer
Sampling Method: Non-Probability Sample
Enrollment: 36 (Estimated)
Dates: Start 2023-10 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Overall survival 2(OS2) | From the date of first fruquinitinib combined with TAS-102 treatment until the date of first documented date of death from any cause , assessed up to 12 months
  Overall survival (OS) of fourth-line treatment of mCRC with fruquinitinib and TAS-102

SECONDARY OUTCOMES:
Objective response rate 2(ORR2, investigator based on RECIST1.1) | from received fruquinitinib combined with TAS-102 to one year
  Objective response rate (ORR) of fourth-line treatment of mCRC with fruquinitinib and TAS-102
Progression-free survival 2(PFS2, investigators based on RECIST1.1) | From the date of first fruquinitinib combined with TAS-102 treatment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 12 months
  Progression-free survival (PFS) of fourth-line treatment of mCRC with fruquinitinib and TAS-102
Disease control rate 2 (DCR2, investigators based on RECIST1.1) | from received fruquinitinib combined with TAS-102 to one year
  Disease control rate (DCR) of fourth-line treatment of mCRC with fruquinitinib and TAS-102

CONTACTS AND LOCATIONS:
Overall Officials: Zhenyu Lin, Principal Investigator — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (3):
- China (3):
  - TONGJI Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Zhongnan Hospital of Wuhan University, Wuhan, Hubei